CLINICAL TRIAL: NCT04261530
Title: Treatment Comparison in Chronic Pain : a Randomized Study
Brief Title: Treatment Comparison in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/85
Record Dates: First submitted 2019-10-21; First posted 2020-02-07 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Comparison of Different Treatment for Chronic Pain
Keywords: Chronic pain; Self-hypnosis; Self-care; Music-therapy; Psycho-education
MeSH Terms: conditions — Chronic Pain | interventions — Self Care

STUDY DESIGN:
Intervention Model Description: Each patients will have a medical consultation and will have to fill-in questionnaires (T0). After, the care staff will have a multidisciplinary discussion and will randomize the participants to different treatment groups : self-hypnosis/self-care, music/self-care, self-care and psycho-education. Another group will be included but will not be randomized because it includes patients who demand to learn self-hypnosis/self-care (group named "self-hypnosis/self-care motivation"). After, participants will receive a 7 months (2 hours session a month) learning program of self-hypnosis/self-care animated by a therapist specialized in hypnosis or music/self-care (identical procedure but the hypnosis is replaced by music) or self-care or psycho-education at the end if which they will complete the same questionnaire (T2). A follow-up at 6 (T3) and 12 (T4) months will also be conducted to account for any long term effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-hypnosis/self-care group (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercice is conducted at the end of each session. A CD with the audiotaped hypnosis exercice is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care
- Music/self-care (Experimental): It is a 7-months 2 hours-session (1 session per month) of music/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. At the end of each session, patients are invited to listen to a relaxing melody of 15 minutes. This melody was composed by a professional musico-therapist. A CD with the audiotaped melody is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Music/self-care
- Self-care (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life.
  Interventions: Behavioral: Self-care
- Psycho-education (Experimental): It is a 7-months 2 hours-session (1 session per month) of psycho-education training. Psycho-education aims to empower and encourage the patient to become an actor in his therapeutic management, while offering a comprehensive model of the mechanisms of pain, the benefits of pharmacological treatments at a physical and psychological level as well as ways to change the way one lives every day.
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Self-hypnosis/self-care
  Arms: Self-hypnosis/self-care group
Behavioral: Music/self-care
  Arms: Music/self-care
Behavioral: Self-care
  Arms: Self-care
Behavioral: Psycho-education
  Arms: Psycho-education

SUMMARY:
Chronic pain concernes one in four adults in Belgium. Because of the psychological and social repercussions, a biopsychosocial approach is necessary in order to improve the quality of life of people suffering from chronic pain. Non-pharmacological techniques such as hypnosis, self-care learning, music-therapy and psycho-education are gaining more and more interest in the scientific field. Indeed, several studies have shown a reduction in psychological distress and an improvement in global quality of life after having learned self-hypnosis/self-care. Furthermore, other studies focusing on music as a treatment for chronic pain highlight an analgesic effect of music over pain and a reduction of common comorbidities. Nevertheless, only few studies aim at comparing these techniques to each other. The aim of our study would be to compare a 7 months learning program of self-hypnosis/self-care, music-therapy/self-care, motivation to learn self-hypnosis/self-care and self-care alone in order to highlight the most efficient treatment for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Fluency in French
* Chronic pain diagnosis

Exclusion Criteria:

* Neurologic disorder
* Psychiatric disorder
* Drug addiction
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Change in pain description | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up))
  The impact of self-hypnosis/self-care on pain description will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (no pain) to 10 (worst pain).
Change in sleep difficulties | T0 (up to 5 month before inclusion), T1 (before the intervention), T2 (up to 8 months)
  The impact of self-hypnosis/self-care upon the severity of insomnia will be assessed by means of the "Insomnia Severity Index" (Morin et al., 2001). Scale ranging from 0 (none) to 4 (very severe).
Change in anxiety | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on anxiety will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in depression | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on depression will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in pain disability | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on pain disability will be assessed by means of the "Pain Disability Index" (PDI, Tait et al., 1990). Scale ranging from 0 (no difficulties) to 10 (a lot of difficulties).
Change in attitudes and beliefs about pain | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the attitudes and beliefs about pain will be assessed my means of the "Survey of Pain Attitudes" (SOPA, Jensen & Karoly, 1987). Scale ranging from 0 (totally wrong) to 10 (totally right).
Change in quality of life | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the quality of life will be assessed by means of the "SF-36"(Ware et al., 1988). Each item is balanced to obtain a score between 0 (worst quality) to 100 (maximum quality).
Change in locus of control | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the locus of control will be assessd my means og the "Multidimensional Health Locus of Control" (MHLC, Wallston et al., 1978). Scale ranging from 1 (no agreement) to 4 (agreement).
Change of the impact of pain | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the impact of pain in individual's life, quality of social support and general activity, will be assessed my means of the "Multidimensional Pain Index" (PDI, Kerns et al., 1985). Scale ranging from 0 (none) to 6 (a lot).
Change in generic health | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on generic health will be assessed by the "EuroQol 5 Dimensions" questionnaire (EQ-5D, Health Policy, 1990). Scale ranging from 1 (no problems) to 3 (extreme problems).
Change in health status | Day 0 (first meeting with the doctor), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of Self-hypnosis/self-care on global health status will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (worst health status) to 100 (best health status).

IPD SHARING:
Plan to Share IPD: No